CLINICAL TRIAL: NCT03020264
Title: Frequency of Hypoglycemia in Patients With Type 2 Diabetes Under Insulin Therapy Older Than 75 Years in Real Life
Acronym: HYPOAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC16_0351
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Type2 Diabetes; Elderly; Hypoglycemia
Keywords: Type 2 Diabetes; Hypoglycemia; Elderly; Insulinotherapy
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients older than 75 years (Experimental): Collection of hypoglycaemia épisodes with the glycemic sensor FREESTYLE Libre Pro
  Interventions: Device: glycemic sensor FREESTYLE Libre Pro

INTERVENTIONS:
Device: glycemic sensor FREESTYLE Libre Pro — Collection of hypoglycemia episodes with glycemic sensor FREESTYLE Libre Pro

SUMMARY:
Diabetes is a chronic and progressive disease that affects nearly 3.5 million people in France.

Currently the investigators are seeing an aging of the population explained by the increase in life expectancy and thus an increasing incidence of diabetes in the elderly. However, the frequency of hypoglycemia in older vulnerable patients remains poorly characterized

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 75 years of age;
* Type 2 diabetes for at least 1 year and treated with insulin for at least 6 months;
* Treated with basal insulin (ie glargine U100: Lantus®, Abasaglar®, glargine U300: Toujeo®, detemir: levemir®, NPH), premix (ie Novomix® and Humalog Mix®), and / Insulin associated or not with one or more oral and / or injectable antidiabetic agents (analog of GLP1...);
* Benefiting from at least 1 capillary glucose per day (carried out by the patient himself or a caregiver);
* Benefiting from a standardized geriatric assessment;
* Signature of informed consent
* Patient benefiting from a social security system.

Exclusion Criteria:

* Male or female aged <75 years;
* Person without diabetes or type 1 diabetes;
* Patient treated only lifestyle modifications and / or oral anti-diabetic drugs and / or GLP-1 receptor agonists alone;
* Subjects with secondary or corticosteroid-induced diabetes;
* Refusal to participate in the study or inability to collect consent;
* Patient for whom follow-up of the study procedures is impossible (glycemic record impossible or insufficient);
* Patient not eligible for geriatric assessment;
* Patient already participating in another study;
* Patient with a severe pathology limiting his life expectancy (palliative care ...) compromising his participation in the study at the discretion of the investigator;
* Patient benefiting from a safeguard of justice.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 161 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Number of confirmed or severe hypoglycemia | 1 month
  Percentage of patients with at least one episode of confirmed and / or severe hypoglycaemia by measuring capillary blood glucose during 4 weeks of prospective follow-up.

SECONDARY OUTCOMES:
number of events / patient / month of severe hypoglycemia | 1 month
  Number of confirmed severe hypoglycaemia episodes (events / patient / month), symptomatic or asymptomatic, occurring in patients during 4 weeks of prospective follow-up.
Number of hospitalizations due to hypoglycemia | 1 month
  Number and duration of hospital stays
Number of asymptomatic confirmed (blood glucose value <0.70g / L) hypoglycemia | 1 month
  Confirmed asymptomatic hypoglycaemia (events / patient / month) occurring in patients collected with the FREESTYLE Libre Pro glucose sensor
Number of hypoglycaemia in elderly patients admitted to EHPAD | 1 month
  Confirmed hypoglycaemia (events / patient / month), symptomatic or asymptomatic, occurring in patients hospitalized in long-term geriatric care sector.
Number of confirmed nocturnal hypoglycaemia (occurring between 0h00-6h00) | 1 month
  Confirmed nocturnal hypoglycaemia (events / patient / month), symptomatic or asymptomatic, occurring in patients
Number of confirmed hypoglycaemia with a threshold blood glucose value <0.54g / L (neuroglucopenic threshold) | 1 month
  Confirmed neuroglucopenic hypoglycaemia (events / patient / month), symptomatic or asymptomatic, occurring in patients
Number of pseudo-hypoglycaemia and unconfirmed hypoglycaemia (Symptoms consistent with hypoglycemia, but with a blood glucose value ≥ 70 mg / dL) | 1 month
  Confirmed pseudo-hypoglycaemia and unconfirmed hypoglycaemia (events / patient / month), occurring in patients
Score for fear of hypoglycemia in elderly diabetic patients | 1 month
  Score for fear of hypoglycaemia (HFS-II)
Number of confirmed and severe hypoglycaemia in patients with type 2 diabetes aged 75 years and older in "vigorous" and "vulnerable" subgroups of patients according to a geriatric assessment score | 1 month
  Confirmed hypoglycaemia (events / patient / month), symptomatic or asymptomatic, occurring in patients
Number of the transition to ER due to hypoglycemia | 1 month
  Number and duration of emergency stays
Number of falls due to hypoglycemia | 1 month
  Number of falls and loss of autonomy (no home support)
Number of death due to hypoglycemia | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CARIOU, Pr, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - CHU de Nantes, Nantes, Loire Atlantique
  - CH d'Ancenis, Ancenis
  - CHU d'Angers, Angers
  - Hôpital Sud Francilien, Corbeil-Essonnes
  - CHRU de Lille, Lille
  - CHU de Poitiers, Poitiers
  - CHU de Toulouse, Toulouse